CLINICAL TRIAL: NCT02035488
Title: Pharmacokinetic Evaluation and Tolerability of Dry Powder Tobramycin by a Novel Device in Patients With Non Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Onno Akkerman, Drs, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tobra-02
Record Dates: First submitted 2013-12-27; First posted 2014-01-14 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Bronchiectasis
Keywords: Dry powder inhalation; Bronchiectasis; Tobramycin
MeSH Terms: conditions — Bronchiectasis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tobramycin (Experimental): Patients with bronchiectasis
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin — Tobramycin dry powder 30 mg inhalation per dose; Dose escalation: 30-60-120 and 240 mg, each one time. One dose per week.
  Other Names: Dry powder tobramycin free base

SUMMARY:
Bronchiectasis is a persistent and frequently progressive condition characterized by dilated and thick-walled bronchi retaining sputum. The main symptoms of bronchiectasis are cough and chronic sputum production. Until now, most patients with non-CF bronchiectasis receive inhaled tobramycin every other month, by use of a nebulizer. However, this delivery system has several disadvantages, like a low lung deposition and pollution with tobramycin in the surrounding environment. With an efficient dry powder inhaler (DPI), a three to six fold higher lung deposition compared to a nebulizer can be obtained. Therapy with a DPI is also less time consuming compared to nebulisation. We will investigate dry powder tobramycin (DP tobramycin) in a novel device in patients with non-CF bronchiectasis. The main objectives of this study are to investigate the pharmacokinetic properties of DP tobramycin at different dosages together with the local tolerability of DP tobramycin via the Cyclops® at different dosages.

DETAILED DESCRIPTION:
Rationale: Bronchiectasis is a persistent and frequently progressive condition characterized by dilated and thick-walled bronchi retaining sputum. The main symptoms of bronchiectasis are cough and chronic sputum production. There is a state of constant colonization with bacteria, which frequently causes exacerbations. The presence of Pseudomonas aeruginosa is an unfavorable prognostic indicator and is associated with increased sputum production, more extensive bronchiectasis on HR-CT of the thorax, more hospitalizations and reduced quality of life. Until now, most patients with non-CF bronchiectasis who are colonized with P. aeruginosa receive inhaled tobramycin every other month, by use of a nebulizer. However, this delivery system has several disadvantages, like a low lung deposition and pollution with tobramycin in the surrounding environment. With an efficient dry powder inhaler (DPI), a three to six fold higher lung deposition compared to a nebulizer can be obtained. Therapy with a DPI is also less time consuming compared to nebulisation. Nebulised tobramycin is used most in routine care; there is also one, rather poorly characterized DPI for tobramycin available, though this DPI is not registrered for non-CF bronchiectasis. We will investigate dry powder tobramycin (DP tobramycin) in a novel device in patients with non-CF bronchiectasis colonized with P. aeruginosa.

Objective: The main objectives are to investigate the pharmacokinetic properties of DP tobramycin at different dosages together with the local tolerability of DP tobramycin via the Cyclops® at different dosages.

Study design: single center, single ascending, single dose, response study. Study population: 8 patients with non-CF bronchiectasis

Main study parameters:

The following pharmacokinetic parameters will be calculated: actual dose (dose minus remainder in inhaler after inhalation), AUC0-12 (area under the curve from 0 -12 h), Cmax (maximum plasma concentration), Tmax (time to maximum plasma concentration), Ka (absorption rate constant), T1/2 el (terminal elimination half-life), CL/F (clearance following pulmonary administration (F= bioavailability)).

Local tolerability of DP tobramycin is determined by scoring adverse events, specifically coughing, and lung function measurement.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants included in this study are patients recruited from the outpatient department of pulmonology. To investigate safety, lung function tests will be performed and the occurrence of adverse events will be scored.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or older
* Obtained informed consent
* Patients having bronchiectasis (confirmed with HR-CT of the chest)

Exclusion criteria:

* Pregnant or breast feeding
* Subjects with known or suspected renal, auditory, vestibular or neuromuscular dysfunction, or with severe, active haemoptysis,
* History of adverse events on previous tobramycin or other aminoglycoside use
* No concurrent use of cyclosporin, cisplatin, amfotericin B, cephalosporins, polymyxins, vancomycin and NSAIDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Actual dose (dose minus remainder in inhaler after inhalation) of tobramycin | one day
Area Under the plasma concentration versus time curve from 0 -12 hours (AUC0-12) of tobramycin •Area Under the plasma concentration versus time curve from 0 -12 hours (AUC0-12) of tobramycin | One day
Maximum plasma concentration (Cmax ) of tobramycin | One day
Time to maximum plasma concentration (Tmax) of tobramycin | One day
Absorption rate constant (Ka) of tobramycin | One day
Terminal elimination half-life (T1/2 el ) of tobramycin | One day
Clearance following pulmonary administration (CL/F) (F= bioavailability) of tobramycin | One day
Decrease of FEV1 in percentage measured by spirometry | One day
Number of Participants with Adverse Events | One day

CONTACTS AND LOCATIONS:
Overall Officials: Huib Kerstjens, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands